CLINICAL TRIAL: NCT01777854
Title: Anti-reflux Control to Decrease Post Tonsillectomy Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patient interest in the study.
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Carissa Wentland DO, DO/Otolaryngology Resident, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GRMC 12 0020
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Laryngopharyngeal Reflux; Throat Pain
MeSH Terms: conditions — Laryngopharyngeal Reflux; Pharyngitis | interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole (Active Comparator): Yes. Omeprazole (generic) will be used. Children >20 kg will be given 20 mg PO daily for 4 weeks prior to tonsillectomy. This is the normal standard pediatric dosing for reflux.
  Omeprazole is authorized to treat reflux in children. The study focuses on laryngopharyngeal reflux that possibly contributes to post tonsillectomy pain.
  Interventions: Drug: Omeprazole
- Sugar pill (Placebo Comparator): The placebo does not look like the omeprazole, however this will not be an issue because none of the subjects will have knowledge of how the medications look.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — The principal investigator will be contacted and will work with the research pharmacist to obtain the omeprazole (20 mg PO daily for patients >20kg) and placebo. The placebo does not look like the omeprazole, however this will not be an issue because none of the subjects will have knowledge of how the medications look. The medication will be locked in the designated medication cabinet at each office. It will be prepackaged for a 28 day course. The patient will start the treatment 4 weeks prior to tonsillectomy and stop the day before surgery. The medication will be given to the patient once the consent and assent are signed. This will avoid an unnecessary office visit to improve patient compliance.
  Other Names: Prilosec, Prilosec OTC

SUMMARY:
The study aims to determine if treating pediatric patients (age 7-17) for four weeks with omeprazole prior to tonsillectomy will decrease post tonsillectomy pain. The hypothesis is that many patients have silent laryngopharyngeal reflux and by reducing the acid entrance into the oropharynx, patients will have less post tonsillectomy pain due to decreased acid irritation of the surgical wound (tonsil fossas).

The study will be a prospective double blind randomized study. Participants will be invited to participate in the study by giving the study information at the preoperative assessment, when the decision is made to have a tonsillectomy performed. If the patient agrees to participate in the study, a written consent and child assent will be obtained and the patient will be randomly assigned to a treatment versus control group based on the randomly assigned participant number.

The treatment group will then be given a four week course of omeprazole to be taken for the four weeks prior to tonsillectomy. The patient will be given a post tonsillectomy assessment form. The form looks at postoperative pain (using a visual analog scale 1-10) as well as oral intake at postoperative day 0,1,3,5,7,10, and 14. The form will be turned in at the postoperative visit or mailed in.

The pain level and oral intake between the two groups to will be compared to determine if antireflux control helps decrease the postoperative pain after tonsillectomy.

DETAILED DESCRIPTION:
The study aims to determine if treating pediatric patients (age 7-18) for four weeks with omeprazole prior to tonsillectomy will decrease post tonsillectomy pain. The hypothesis is that many patients have silent laryngopharyngeal reflux and by reducing the acid entrance into the oropharynx, patients will have less post tonsillectomy pain due to decreased acid irritation of the surgical wound (tonsil fossas).

The study will be a prospective double blind randomized study. Participants will be invited to participate in the study by giving the study information at the preoperative assessment, when the decision is made to have a tonsillectomy performed. If the patient agrees to participate in the study, a written consent and child assent will be obtained and the patient will be randomly assigned to a treatment versus control group based on the randomly assigned participant number.

The treatment group will then be given a four week course of omeprazole or placebo to be taken for the four weeks prior to tonsillectomy. The investigators will be blinded to the intervention. The medication will be kept in a locked drawer at the ENT Associates office. The patient will take the medication 20 mg orally once a day for 28 days prior to the procedure with day 28 being the day before the tonsillectomy. The patient will be provided with a calender that is marked with the start date of the medication. The patient is to document any missed doses on the calender. On the day of surgery, the patient will return the remainder of the medication in an opaque bag along with the calender and this will be given back to the research pharmacist to account for the medication.

The patient will be given a post tonsillectomy assessment form. The form looks at postoperative pain (using a visual analog scale 1-10) as well as oral intake at postoperative day 0,1,3,5,7,10, and 14. The form will be turned in at the postoperative visit (2 weeks after the surgery) or mailed in.

The pain level and oral intake between the two groups to will be compared to determine if antireflux control helps decrease the postoperative pain after tonsillectomy.

Other variables collected will be patient age, gender, method of surgery, pain medication prescribed, and indication for procedure. The data will be stored in a password protected computer files and the patient will only be identified by study number.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-17 years old
* Weight >20 kg
* Scheduled to undergo a tonsillectomy (with or without adenoidectomy) in greater than four weeks.
* Health conditions (any of the following): Hypertrophic tonsils and adenoids, sleep disordered breathing, obstructive sleep apnea, chronic or recurrent tonsillitis, halitosis, dysphagia
* Must be able to swallow pills or tolerate taking the medication sprinkled on applesauce or other soft food.

Exclusion Criteria:

* Age <7
* Weight <20kg
* Patients declared by the parent not able to communicate pain level.
* Patients whose tonsillectomy is scheduled <4 weeks from the preoperative assessment (The patient would not have time to complete the preoperative treatment) (An exception to this exclusion criteria will be for the control group)
* Patients with a mental illness. This will be determined by the patient's physician or the physician overseeing the care of the patient.
* Unable to swallow pills or tolerate sprinkling the medication on soft food.
* Pregnant patients
* Any patients already taking Proton Pump Inhibitor

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carissa J Wentland, DO, Principal Investigator — Ascension Health; Kimberly Barber, PhD, Study Director — Ascension Health; Candy Rainwater, Study Director — Ascension Health
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Omeprazole: Omeprazole (generic) will be used. Children >20 kg will be given 20 mg PO daily for 4 weeks prior to tonsillectomy. This is the normal standard pediatric dosing for reflux.
  Omeprazole is authorized to treat reflux in children. The study focuses on laryngopharyngeal reflux that possibly contributes to post tonsillectomy pain.
  Omeprazole: The principal investigator will be contacted and will work with the research pharmacist to obtain the omeprazole (20 mg PO daily for patients >20kg) and placebo. The placebo does not look like the omeprazole, however this will not be an issue because none of the subjects will have knowledge of how the medications look. The medication will be locked in the designated medication cabinet at each office. It will be prepackaged for a 28 day course. The patient will start the treatment 4 weeks prior to tonsillectomy and stop the day before surgery. The medication will be given to the patient once the consent and assent are signed. This will avoid an
Period: Overall Study
Arm/Group | Omeprazole | Sugar Pill
Started (Study was terminated before patients had intervention.) | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Pre Treatment: the study was terminated before patients received the medication The study did not progress to the point where the patients were randomized into different arms.
Arm/Group | Pre Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants] — between 7 and 18
  Participants
    <=18 years | 6
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 14 [7 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Pain After Tonsillectomy
Description: A questionnaire will be given to patients. Patients are asked to describe their pain and oral intake on post op days 0,1,3,5,7,10 and 14. This should take less than one minute per assessment day. At the end of the survey, they are asked to comment on any postoperative problems such as hemorrhage or dehydration. This should take less than 5 minutes. Parents will be asked to assist the child in completing the survey. They will be asked to turn in the form on the postoperative follow up visit (14-21 days after surgery) or mail it in to the principal investigator if the surgeon does not have a postoperative follow up visit. For these patients, an addressed and stamped envelope will be provided.
Time Frame: 2 weeks
Population: The patients did not receive the intervention
Arm/Group | Pre Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The data was not collected.
Description: This data was not collected.
Groups:
- Pre Treatment: This data was not collected
Arm/Group | Pre Treatment
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No